CLINICAL TRIAL: NCT05792787
Title: Association Between Apical Periodontitis and Atherosclerotic Cardiovascular Diseases: a Case-control Study
Brief Title: Association Between Apical Periodontitis and Atherosclerotic Cardiovascular Diseases
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Simone Grandini, Professor, University of Siena
Other Study IDs: CVD001
Record Dates: First submitted 2023-02-16; First posted 2023-03-31 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Apical Periodontitis; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Periapical Periodontitis; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Apical Periodontitis: Patients with radiographic signs of Apical Periodontitis. The inclusion criteria of the study are healthy patients older than 40 years old, the presence of at least 24 teeth and the ability and willingness to give informed consent. Participants affected by any systemic disease or being administered either antibiotics in the last 6 months or antiaggregant, antiplatelet and antihypertensive medications are excluded from this study.
  The atherosclerosis risk factors excluded in our study are signs of CVD, smoking habits, diabetes , obesity, arterial hypertension, dyslipidemia. Patients with periodontal disease and lesions other than endodontic etiology in maxilla/mandible will be also excluded from this study ). Participants that were pregnant or lactating females, non-Italian or only English speaking will also also excluded from the study, as well as those who were unable or unwilling to give informed consent.
  Interventions: Diagnostic Test: Echo-color-doppler
- Control: healthy individual free from clinical and radiographic evidence of AP. The inclusion criteria of the study are healthy patients older than 40 years old, the presence of at least 24 teeth and the ability and willingness to give informed consent. Participants affected by any systemic disease or being administered either antibiotics in the last 6 months or antiaggregant, antiplatelet and antihypertensive medications are excluded from this study.
  The atherosclerosis risk factors excluded in our study are signs of CVD, smoking habits, diabetes , obesity, arterial hypertension, dyslipidemia. Patients with periodontal disease and lesions other than endodontic etiology in maxilla/mandible will be also excluded from this study ). Participants that were pregnant or lactating females, non-Italian or only English speaking will also also excluded from the study, as well as those who were unable or unwilling to give informed consent.
  Interventions: Diagnostic Test: Echo-color-doppler

INTERVENTIONS:
Diagnostic Test: Echo-color-doppler — To perform the initial screening patients will undergo panoramic radiography and clinical examination followed by periapical radiographs of the teeth suspected of AP using the long cone paralleling technique with a film holder. The following parameters will be recorded:
  1. The number of decayed, missing and filled teeth (DMFT index)
  2. The number of teeth with AP
  3. Periapical Index Score All individuals will undergo a cardiovascular examination in the Unit of Vascular Surgery, University of Siena (Siena, Italy). The cardiovascular assessment included physical examination, blood pressure measurement, past medical history and echo-color-doppler for the assessment of carotid intima-media thickness (cIMT), presence of abdominal aortic aneurysm and presence of peripheral pulses.
  Other Names: Cardiovascular Examination

SUMMARY:
The aim of the study is to evaluate the association between apical periodontitis (AP) and atherosclerotic cardiovascular disease (ASCVD) by assessing the multiplicative effect of AP on secondary outcomes of ASCVD. Sixty-two subjects will be enrolled from the Unit of Endodontics and Restorative dentistry and allocated into 2 distinct groups depending on the presence or absence of periapical lesions. Group 1 will be composed of 31 patients with radiographic signs of AP. On the contrary, another 31 healthy individual (free from clinical and radiographic evidence of AP) meeting the inclusion and exclusion criteria were included as controls (group 2) A complete dental examination will performed on each patient in both groups. All the patients will be subjected to a cardiovascular examination to assess carotid intima-media thickness (cIMT), presence of abdominal aortic aneurysm, presence of peripheral pulses through echo-color-doppler.

DETAILED DESCRIPTION:
The aim of the present case-control study is to evaluate the multiplicative effect of AP on secondary outcomes of ASCVD. Sixty-two subjects will be enrolled from the Unit of Endodontics and Restorative dentistry of the university of Siena.

The inclusion criteria of the study are healthy patients older than 40 years old, the presence of at least 24 teeth and the ability and willingness to give informed consent.Participants affected by any systemic disease or being administered either antibiotics in the last 6 months or antiaggregant, antiplatelet and antihypertensive medications will be excluded from this study.

The atherosclerosis risk factors excluded in our study are prior or existing signs of CVD, smoking habits, diabetes, obesity, arterial hypertension, dyslipidemia, and echocardiographically detectable left ventricular hypertrophy. Patients with periodontal disease and lesions other than endodontic etiology in maxilla/mandible are also excluded from this study. Participants that were pregnant or lactating females, non-Italian, or only English-speaking are also excluded from the study, as well as those who were unable or unwilling to give informed consent.

Sixty-two subjects fulfilling the previously described criteria will be enrolled from the outpatient department and allocated into two distinct groups depending on the presence or absence of periapical lesions. Group 1 will be composed of 31 patients with radiographic signs of AP. On the contrary, another 31 healthy individuals (free from clinical and radiographic evidence of AP) meeting the inclusion and exclusion criteria will be included as controls (group 2) and matched on age, BMI, sex, and physical characteristics. AP cases will be designated those patients with at least one tooth exhibiting radiographic evidence of apical radiolucency exceedingly twice the width of the periodontal ligament space. A complete dental examination will be performed on each patient in both groups.

To perform the initial screening, patients will undergo panoramic radiography and clinical examination followed by periapical radiographs of the teeth suspected of AP using the long cone paralleling technique with a film holder. The following parameters will be recorded:

1. The number of decayed, missing, and filled teeth (DMFT index)
2. The number of teeth with AP
3. Periapical Index Score All measurements will be recorded by one endodontist (GM). All individuals will undergo cardiovascular examination in the Unit of Vascular Surgery, University of Siena (Siena, Italy). The cardiovascular assessment included physical examination, blood pressure measurement, past medical history, and echo-color-doppler where carotid intima-media thickness (cIMT), presence of abdominal aortic aneurysm, presence of peripheral pulses through echo-color-doppler will b assessed.

The results expected from this study are:

* a significant increase in ASCVD secondary parameters (outcomes) in patients with PA (exposure factor), compared with subjects without PA;
* significant association between BP and the presence of peripheral pulses and abdominal aortic aneurysm, respectively.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 40 years old
* the presence of at least 24 teeth
* the ability and willingness to give informed consent

Exclusion Criteria:

* any systemic diseases
* antibiotic administration in the last 6 months
* antiaggregant, antiplatelet and antihypertensive medications
* existing signs of CVD
* smoking habits, diabetes
* obesity
* arterial hypertension
* dyslipidemia
* periodontal disease
* lesions other than endodontic etiology in maxilla/mandible were also excluded from this study
* pregnant or lactating females non-Italian or only English speaking
* inability or unwillingness to give informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty-two subjects fulfilling the previously described criteria will be allocated into 2 distinct groups depending on the presence or absence of periapical lesions. Group 1 will be composed of 31 patients with radiographic signs of AP. On the contrary, another 31 healthy individual (free from clinical and radiographic evidence of AP) meeting the inclusion and exclusion criteria will be included as controls (group 2) and matched on age, BMI, sex and physical characteristics. AP cases will be designated as those patients with at least 1 tooth exhibiting radiographic evidence of apical radiolucency exceedingly twice the width of the periodontal ligament space.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Carotid Intima medial Thickness (c-IMT) | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  C-IMT measurements are done in mm, and they are taken from the right and left common carotid artery (CCA) and they are used as surrogate endpoints to diagnose early signs of carotid atherosclerotic cardiovascular diseases.
Presence of Carotid Plaque | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  the presence of atherosclerotic plaques is considered as a surrogate endpoint point variable to diagnose early alterations of carotid atherosclerotic cardiovascular disease. Plaque is defined as a focal structure that encroaches into the arterial lumen of at least 0.5 mm or 50% of the surrounding IMT value or demonstrates a thickness >1.5 mm as measured from the media-adventitia interface to the intima-lumen interface.

SECONDARY OUTCOMES:
North American Symptomatic Carotid Endarterectomy Trial (NASCET) | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  The NASCET method is used to calculate the percentage of stenosis in carotid arteries. The NASCET percentage is the ratio between the residual diameter at the stenosis and the surface of the distal normal lumen where there is no stenosis subtracted by the residual diameter at the stenosis.
Ankle Brachial Index (ABI) | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  The ankle-brachial index (ABI) is a non-invasive tool for the assessment of vascular status. It consists of the ratio between the systolic blood pressure of the lower extremity (i.e., the ankle) and the upper extremity.
Right and Left Common Iliac Arteries (CIA) diameter | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  Measuring the diameter of the CIAs (mm) can be done to assess for potential conditions such as peripheral artery disease (PAD) or an abdominal aortic aneurysm (AAA
Abdominal aorta maximum diameter | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  Measuring the diameter of the abdominal aorta (mm) can be done to assess for potential abdominal aortic aneurism.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Grandini, PhD, DDS, Principal Investigator — University of Siena
Locations (1):
- Azienda Ospedaliera Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: Undecided